CLINICAL TRIAL: NCT00324441
Title: A Randomized Controlled Trial on the Effectiveness of Mild Water-Filtered Near Infrared Hyperthermia as an Adjunct to a Standard Multimodal Rehabilitation in the Treatment of Fibromyalgia
Brief Title: Mild Water-Filtered Near Infrared Whole-Body-Hyperthermia as an Adjunct in the Treatment of Fibromyalgia
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Forschungsinstitut für Balneologie und Kurortwissenschaft Bad Elster (Other Government)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: WBH-FM-1
Record Dates: First submitted 2006-05-09; First posted 2006-05-11 (Estimated); Last update posted 2006-05-11 (Estimated); Status verified 2003-08

CONDITIONS: Fibromyalgia
Keywords: Fibromyalgia; Rehabilitation; Physical Medicine; Whole-Body Hyperthermia; Water-Filtered Near Infrared
MeSH Terms: conditions — Fibromyalgia

INTERVENTIONS:
Device: Iratherm® 1000

SUMMARY:
The purpose of the study is to evaluate whether mild walter-filtered near infrared hyperthermia produces an additional benefit when applied as an adjunct to standard multimodal rehabilitation compared to standard multimodal rehabilitation only in patients with fibromyalgia.

DETAILED DESCRIPTION:
Mild systemic heat agents, including infrared whole-body hyperthermia, are used as treatment options in multimodal rehabilitation programs for fibromyalgia in Germany. However, no randomized controlled clinical trial exists on their effectiveness for this condition.

This study is designed as an add-on study to evaluate the additional benefit of mild walter-filtered near infrared hyperthermia and a standard multimodal rehabilitation program compared to a standard multimodal rehabilitation program only. Standard multimodal rehabilitation is configured as usually applied in clinical trials with exercise, cognitive behavioral therapy, and health education as the main treatment components.

Mild walter-filtered near infrared hyperthermia (heating-up to 38.1 degrees C body core temperature followed by a 15-min heat retention period) is administered twice a week over 3 weeks during a rehabilitation hospital stay.

Primary outcome measures are measured at baseline, postintervention, 3 and 6 months postintervention. Analysis is done by intention to treat, for significance testing Repeated Measures ANCOVA is used.

ELIGIBILITY:
Inclusion Criteria:

* participants must meet the American College of Rheumatology 1990 criteria for fibromyalgia
* participants must report a score ≥ 4 on the pain intensity subscale of the Fibromyalgia Impact Questionnaire (range: 0-10)
* participants must report a score ≥ 4 on the normalized physical functioning subscale of the Fibromyalgia Impact Questionnaire (range: 0-10)
* participants must be aged between 18 and 70 years

Exclusion Criteria:

* severe cardiovascular disease
* metabolic disease
* nervous system disorder
* blood coagulation disease
* cancer
* acute inflammatory disease
* status after organ transplantation
* reduced general health (Karnofsky Index ≤ 50)
* pregnant women
* breast feeding women
* persons involved in a pending litigation for early pensioning due to fibromyalgia
* persons planning to apply for a pension due to fibromyalgia

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 132
Dates: Start 2004-01; Study Completion 2005-07

PRIMARY OUTCOMES:
affective pain (German version of the McGill Pain Questionnaire)
sensory pain (German version of the McGill Pain Questionnaire)

SECONDARY OUTCOMES:
pain intensity (visual analogue scale)
Fibromyalgia related quality of life(German version of the Fibromyalgia Impact Questionnaire)
tender point assessment(mean tender point pain threshold, total tender point intensity, tender point count)
adverse events, side effects

CONTACTS AND LOCATIONS:
Overall Officials: Thomas Brockow, MD, Study Chair — FBK Bad Elster
Locations (1):
- Rehabilitationsklinik Hoher Meissner, Bad Sooden-Allendorf, Hesse, Germany